CLINICAL TRIAL: NCT06437587
Title: Effects of Appropriate Technology for Home-based Rehabilitation in Patients With Post-stroke Physical Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xi Chen (Other)
Collaborators: Harbin Medical University (Other)
Responsible Party: Sponsor-Investigator, Xi Chen, researcher, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HMUDQ20231116205
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Stroke
Keywords: home-based rehabilitation; appropriate technology
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the nature of the intervention, it is impossible to blind the researcher of the intervention who will deliver the intervention. Therefore, the participants and the outcome assessor will be blinded. The outcome assessor will be blinded to the allocation throughout the study and will independently assess all outcomes at T0, T1, and T2 for both groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Home-based rehabilitation appropriate technology (S-HRAT) training
  Interventions: Other: Home-based rehabilitation appropriate technology (S-HRAT) training
- control group (No Intervention): Routine discharge instructions

INTERVENTIONS:
Other: Home-based rehabilitation appropriate technology (S-HRAT) training — The S-HRAT training instruction consists of two phases: in-hospital training and post-discharge remote home training. Based on the S-HRAT list, we select individualized home rehabilitation training exercises for the participants and conduct five offline training instruction sessions one week before discharge to ensure that the participants master the correct method for each exercise and clarify precautions. At discharge, participants will receive an S-HRAT brochures, which will include detailed text, pictures and video demonstrations of exercises, to visualize the rehabilitation instructions and make them easy to understand. Participants learn how to use the S-HRAT booklet and follow a daily training program to complete the prescribed content. They will be asked to record a video of their training and send it to the researcher via WeChat for monitoring purposes and feedback.
  Arms: intervention group

SUMMARY:
The goal of this clinical trial is to assess the effect of S-HRAT to improve patients' motor function and activities of daily living.

DETAILED DESCRIPTION:
Limb dysfunction is the primary disability factor among stroke patients. However, due to various factors, most stroke survivors do not receive sufficient rehabilitation training after discharge. Home-based rehabilitation appropriate technology (S-HRAT） training could be a strategy to meet the patients' requirements for rehabilitation after hospital discharge. This study aims to assess the effect of a nursing intervention based on Cox's Interaction Model of Client Health Behavior (IMCHB) with the application of S-HRAT to improve patients' motor function and activities of daily living.

In this pilot trial, 36 stroke survivors with limb dysfunction will be screened for inclusion before hospital discharge and randomly assigned to the experimental or control group with their informed consent. The control group(n=18) will receive the usual care provided by the hospital. The experimental group(n=18) will receive usual care and an 8-week S-HRAT training program. This nursing interventions use Cox's IMCHB as a theoretical framework that consists of rehabilitation exercises and the provision of health information. Baseline assessments will be conducted on the day before hospital discharge, and outcomes will be assessed at 8 weeks and 12 weeks after discharge. The primary outcome is change in motor function 8 weeks after discharge, and the secondary outcomes include the activities of daily living, anxiety, depression, exercise adherence, and patient satisfaction.

This study is the first of its kind conducted in China to use Cox's IMCHB as a framework to guide the development of the S-HRAT training program. Our pilot will determine if such an approach is feasible and effective in enhancing motor function and improving the activities of daily living post-stroke after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18;
* Patients diagnosed with cerebrovascular disease who have cerebral infarction or cerebral hemorrhage based on cranial CT or MRI and meet the diagnostic criteria;
* Patients are in the non-acute phase, meaning between two weeks and six months after the onset of the disease;
* Patients with limb dysfunction.

Exclusion Criteria:

* Return to a hospital or rehabilitation facility after discharge;
* The patient has a history of mental illness and dyslexia;
* Patients have a combination of serious, life-threatening conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Motor Function | baseline (T0), 8-week post-intervention (T1), and 12-week follow-up (T2).
  The motor function of the patients is measured using the Motor Assessment Scale (MAS) for stroke. MAS is methodologically simple, targeted, and easily generalizable for motor function assessment in stroke patients, as well as reliable and valid. The scale consists of nine items, each of which is scored from 0 to 6 out of 48, with the ninth item not scoring. Higher scores indicate better motor function.
Balance | baseline (T0), 8-week post-intervention (T1), and 12-week follow-up (T2).
  Balance was measured using the Berg Balance Scale (BBS). The scale consists of 14 items, including sitting to standing, standing independently, walking independently, and standing to sit, and each item is scored on five functional levels: 0, 1, 2, 3, and 4. A score of 4 indicates that the action under examination can be performed normally. In contrast, a score of 0 indicates that it cannot be performed or requires significant assistance. The total possible score is 56, with higher scores indicating better balance.

SECONDARY OUTCOMES:
Activity of Daily Living | baseline (T0), 8-week post-intervention (T1), and 12-week follow-up (T2).
  The Modified Barthel Index(MBI) is used to measure the activity of daily living. The scale consists of ten items, including eating, bathing, grooming, dressing, toileting, bed and chair transfers, walking on level ground, walking up and downstairs, bowel control, and urinary control. The possible score ranges from 0 to 100, and a higher score means greater independence
Exercise Adherence | baseline (T0), 8-week post-intervention (T1), and 12-week follow-up (T2).
  The Functional Exercise Adherence Scale for Stroke Patients (questionnaire of exercise adherence, EAQ) developed by Chinese author Beilei Lin in 2013 was used to assess patients' adherence to rehabilitation exercises. The scale consists of three dimensions: physical participation in exercise, monitoring of exercise effects, and active adherence to seeking exercise advice. Each item is scored using a Likert scale ranging from 0 to 4, with a total score ranging from 14 to 56. A higher score indicates a higher level of exercise adherence.
Patient Satisfaction | baseline (T0), 8-week post-intervention (T1), and 12-week follow-up (T2).
  The Nursing Job Satisfaction Questionnaire (Client Satisfaction Test, CST) was developed by Bear Bowers based on the IMCHB model and comprises 12 items across six domains: emotional support, health information, decision control, professional skills, service accessibility, and overall satisfaction. The rating method employs a scale of 1 to 5 points, representing five options "very satisfied," "quite satisfied," "not sure," "not too satisfied," and "very dissatisfied." The total scale thus ranges from 12 to 60 points. A higher score on the scale indicates a higher level of patient satisfaction.
Anxiety and Depression | baseline (T0), 8-week post-intervention (T1), and 12-week follow-up (T2).
  The Chinese version of the Hospital Anxiety and Depression Scale (HADS) is employed to assess the anxiety and depression levels of patients. The HADS is a frequently used instrument for assessing the severity of anxiety and depression in patients. It is a 14-item instrument comprising two subscales: anxiety (HADS-A, 7 items) and depression (HADS-D, 7 items). Each item is rated on a 4-point Likert scale, ranging from 0 for "no problem" to 3 for "severe problem," with higher scores indicating higher levels of anxiety and depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Daqing Oilfield General Hospital, Daqing, Heilongjiang, China